CLINICAL TRIAL: NCT04702841
Title: Clinical Application of Chimeric Antigen Receptor Modified γδ T Cells（CAR - γ δ T Cells） in Relapsed and Refractory CD7 Positive T Cell-derived Malignant Tumors
Brief Title: CAR - γ δ T Cells in the Treatment of Relapsed and Refractory CD7 Positive T Cell-derived Malignant Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-ky012
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: CAR; Malignant Tumors
Keywords: CD7 Positive T-cell; γδT
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-γδT (Experimental): Infusion,iv,0.2-5 ×10^6/ kg,once.
  Interventions: Drug: Chimeric antigen receptor modified γδ T cells

INTERVENTIONS:
Drug: Chimeric antigen receptor modified γδ T cells — Dosage: the total dosage of reinfusion is 0.2-5 × 10^6 / kg, which is determined according to the body weight of the subject and the effective content of cell preparation.
  Other Names: CAR-γδT cell infusion

SUMMARY:
This is a study on the clinical application of chimeric antigen receptor modified γδ T cells (CAR - γδ T cells) in relapsed and refractory CD7 Positive T cell-derived malignant tumors.The main purpose of this study was to evaluate the efficacy of car - γ δ T cell infusion in patients with relapsed and refractory CD7 Positive T cell-derived malignancies.

DETAILED DESCRIPTION:
γδT cells are known as "a great candidate for car-t cells". Although they only account for 2% - 5% of all T cells in our body, they are a natural killer.

CD7 is recognized as a sensitive marker of T-ALL, and its expression level on T-ALL cells is opposite to CD3: compared with normal T cells, the expression level of CD7 on T-ALL cells is significantly increased (P < 0.001), while the expression level of CD3 on T-ALL cells is significantly decreased (P < 0.001). At the same time, CD7 expression is absent in about 10% of normal T cells, and these CD7 negative T cells have the ability of normal T cells to express cytokines. Therefore, CD7 has become a potential target for the treatment of T-ALL because of its specificity and safety.

ELIGIBILITY:
Inclusion Criteria:

1. the patients must be patients with relapsed or refractory CD7 Positive T cell-derived malignancies, who have at least one course of standard regimen chemotherapy and one course of salvage regimen chemotherapy and have poor effect;
2. Researchers believe that there is no other feasible and effective alternative treatment, such as hematopoietic stem cell transplantation;
3. Patients should have indicators for detection or evaluation of disease, including detection of minimal residual disease (MRD) by immunophenotyping, cytogenetics or PCR;
4. They are 14-70 years old, regardless of gender or race;
5. Physical condition: ECoG score 0-2;
6. Cardiac function: left ventricular ejection fraction greater than or equal to 40%;
7. The expected survival time was > 12 weeks;
8. Serum creatinine (CR) ≤ 1.5 × ULN (upper limit of normal value), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, total bilirubin ≤ 1.5 × ULN;
9. Patients have self-knowledge ability and can sign informed consent;
10. The guardian of the child patient agreed to sign the informed consent.

Exclusion Criteria:

1. pregnant or lactating women;
2. Uncontrolled infection;
3. Active HBV or HCV infection;
4. People living with HIV;
5. Less than 100 days after allogeneic hematopoietic stem cell transplantation;
6. Patients with acute GVHD or chronic GVHD after allogeneic hematopoietic transplantation;
7. Patients receiving GVHD treatment.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
ORR 3 | three months after CAR-T cells infusion
  3-month objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Xingbing Wang, Principal Investigator — No.1, Swan Lake Road, new administrative and Cultural District, Hefei City, Anhui Province
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China